CLINICAL TRIAL: NCT01813942
Title: Platform for Medical Information Extraction From Incomplete Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201302013RINC
Record Dates: First submitted 2013-03-05; First posted 2013-03-19 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Liver Cancer
Keywords: clinical narrative report; time series data; missing value
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In order to perform research smoothly, the process of information extraction is required for translating data in clinical text into available format for analysis and statistic. In medical research, the problem of missing data occurs frequently. It is important to develop the method with better imputation performance in the stability and accuracy. The purposes of this project are to provide the data integration and extraction methods for handling the structured and unstructured data sources in more efficient ways, to provide the validation scheme for facilitating the data reviewing of extracted results produced by information extraction modules, to increase the quality of clinical data by comparing the data from different data sources and correcting data errors and inconsistent, to handle the clinical data with the properties of time series and incompleteness, to increase accuracy of data analysis and increase quality of health care by improving the completeness and correctness of clinical data, to provide flexibility of methods in the platform. In the project, the disease topic is focused on the liver cancer patients' clinical data and we hope the methods in the projects can be extended to handle other diseases by replacing these knowledge models in the future.

DETAILED DESCRIPTION:
Because of the increasing adoption of Electronic Medical Record (EMR) systems, the data access of EMR is more and more convenient. However, there still have difficulties in analyzing all the clinical data directly due to a large number of records using the narrative format. In order to perform research smoothly, the process of information extraction is required for translating data in clinical text into available format for analysis and statistic. In medical research, the problem of missing data occurs frequently. It is important to develop the method with better imputation performance in the stability and accuracy. The purposes of this project are to provide the data integration and extraction methods for handling the structured and unstructured data sources in more efficient ways, to provide the validation scheme for facilitating the data reviewing of extracted results produced by information extraction modules, to increase the quality of clinical data by comparing the data from different data sources and correcting data errors and inconsistent, to handle the clinical data with the properties of time series and incompleteness, to increase accuracy of data analysis and increase quality of health care by improving the completeness and correctness of clinical data, to provide flexibility of methods in the platform. In the project, the disease topic is focused on the liver cancer patients' clinical data and we hope the methods in the projects can be extended to handle other diseases by replacing these knowledge models in the future.

ELIGIBILITY:
Patients with liver cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The number of patients correctly identified by recurrence predictive model | 3 years
  The recurrence predictive model is developed using the incomplete data set, this model is used for predicting the recurrent status of patient who received the specific treatment for liver cancer. The number of patients correctly identified by recurrence predictive model is regarded as the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Feipei Lai, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan